CLINICAL TRIAL: NCT06036329
Title: Evaluating the Usability and Performance of a PAP Mask System in the Home Environment
Brief Title: Whitsundays (Nasal) Mask Take Home Study (90 Days)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SLP-23-02-01; D638-1118 (Other: ResMed)
Record Dates: First submitted 2023-07-18; First posted 2023-09-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group A provided with 1 Whitsundays Nasal mask without a spare mask cushion (Experimental): • Provided with 1 Whitsundays Nasal mask without a spare mask cushion (To be provided as requested)
  Interventions: Device: Group A : provided with 1 Whitsundays Nasal mask without a spare mask cushion
- Group B provided with 1 Whitsundays Nasal mask with 2 spare mask cushions (Experimental): • Provided with 1 Whitsundays Nasal mask with 2 spare mask cushions
  Interventions: Device: Group B : provided with 1 Whitsundays Nasal mask with 2 spare mask cushions

INTERVENTIONS:
Device: Group A : provided with 1 Whitsundays Nasal mask without a spare mask cushion — Group A will be provided with 1 Whitsundays Nasal mask without a spare mask cushion (replacement cushions will only be provided when requested)
  Arms: Group A provided with 1 Whitsundays Nasal mask without a spare mask cushion
Device: Group B : provided with 1 Whitsundays Nasal mask with 2 spare mask cushions — Group B will be provided with 1 Whitsundays Nasal mask with 2 spare mask cushions
  Arms: Group B provided with 1 Whitsundays Nasal mask with 2 spare mask cushions

SUMMARY:
The goal of this multi-site, prospective, randomized, double arm study without blinding is to test the usability of the Whitsundays mask system at home by patients with Obstructive Sleep Apnea. The main questions it aims to answer are:

* How the Whitsundays masks performs in the home environment
* What is the subject's first impression of the Whitsundays mask and what is their preference compared to their own mask
* What is the difference between the subject's objective therapy data when using the Whitsundays mask compared to their own mask
* Is there wear and tear of the Whitsundays mask and how frequently do the cushions need replacement Participants will be asked to use the Whitsundays mask for 90 days, answer questionnaires about the initial impression of the mask, the performance of the mask, and their preference compared to their own mask. Researchers will compare one group of subjects who will be provided with cushion replacements to another group who will only be provided with cushion replacements upon request to determine the need for cushion replacement, its frequency, and the reasons for cushion replacement during home usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients who ≥ 18 years of age
* Patients being treated for OSA with a PAP device for ≥ 6 months
* Patients currently using a ResMed PAP device (S9, AirSense 10 & AirSense 11) compatible with AirView (with cellular data connectivity and has been sending device data to the cloud)
* Patients currently using ResMed AirFit N30i or Philips DreamWear™ Nasal
* Patients who are willing to try the prototype mask for up to 90 nights
* Patients who are willing to take photos of the prototype mask every 2 weeks for the duration of the study
* Patients who reside in the USA and intend to stay in the USA for the next 6 months
* Patients with access to the internet (such as a smartphone or laptop) to complete online surveys

Exclusion Criteria:

* Patients using Bilevel flow generators
* Patients who are or may be pregnant
* Patients with a preexisting lung disease/condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* If you are pregnant or planning to become pregnant
* Patients believed to be unsuitable for inclusion by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
11 point Likert Scale Questionnaire | 90 days
  • Subjective scores will be collected from subjects on each attribute being assessed (e.g. visual appeal, ease of use, ease of cleaning, seal, comfort, overall performance etc.). Scores will be collected using an 11-point Likert Scale Questionnaire. Minimum value will be zero. Maximum value will be 10. A higher score indicates better outcomes. A score of 10 is considered very favorable, and a score of 0 is very unfavorable.

SECONDARY OUTCOMES:
11 point Likert Scale Questionnaire | 90 days
  • Subject's subjective impression and comments comparing the prototype mask (Whitsundays Nasal) to the subject's current mask with regards to ease of use, visual appearance, seal, comfort, facial markings, noise and overall performance. • Scores will be collected using an 11-point Likert Scale Questionnaire. Minimum value will be zero. Maximum value will be 10. A higher score indicates better outcomes. A score of 10 is considered very favorable, and a score of 0 is very unfavorable.
Apnea Hypopnea Index (AHI) | 90 days
  • The AHI recorded by the subject's PAP device while using their own mask will be compared to the AHI recorded by the subject's PAP device while using the Whitsundays mask. The AHI will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.
Compliance | 90 days
  • The subject's average daily hours of use of PAP therapy recorded by the subject's PAP device while using their own mask will be compared to the average daily hours of use recorded by the subject's PAP device while using the Whitsundays mask. The average daily hours of use will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.
Leak | 90 days
  The median air leak (L/minute) recorded by the subject's PAP device while using their own mask will be compared to the median air leak (L/minute) recorded by the subject's PAP device while using the Whitsundays mask. The median air leak will be obtained from the ResMed AirView Compliance Reports downloaded during the study visits.
Pressure Differences | 90 days
  The median air pressure (cmH2O) used during PAP therapy recorded by the subject's PAP device while using their own mask will be compared to the median air pressure (cmH2O) recorded by the subject's PAP device while using the Whitsundays mask. The median air pressure levels will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.
Frequency of Cushion Replacement | 90 days
  • Subject's frequency of cushion replacement will be recorded using the Mask Cushion Change Form to be provided to Group B participants on Day 14 and every 2 weeks for the duration of the study. The Mask Cushion Change form will be provided to Group A participants who request a cushion change.
Reason for Cushion Replacement | 90 days
  • Subject's reason for cushion replacement will be recorded using the Mask Cushion Change Form to be provided to Group B participants on Day 14 and every 2 weeks for the duration of the study. The Mask Cushion Change form will be provided to Group A participants who request a cushion change.
Deterioration of Mask | 90 days
  • Photos of the subject's prototype mask system taken at 2-week intervals to observe any visual deterioration such as cracking, crazing, tears, dirt or stain build up

CONTACTS AND LOCATIONS:
Overall Officials: William Hevener, RPSGT, Principal Investigator — Sleep Data; Matthew Uhles, MS, Principal Investigator — Clayton Sleep Institute
Locations (2):
- United States (2):
  - Sleep Data, San Diego, California
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No